CLINICAL TRIAL: NCT05061576
Title: Instructed Home-based Physical Exercise for Patients With Liver Cirrhosis
Acronym: INSPEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Hannes Hagström, Principal Investigator, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-04454
Record Dates: First submitted 2021-09-09; First posted 2021-09-29 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Oral advice on exercise from a physician.
  Interventions: Behavioral: Standard of Care advice on physical activity
- Active intervention (Experimental): A leaflet with instructions and images on different forms of physical activities as well as clear recommendations on when to perform these.
  Interventions: Behavioral: Structured advice on physical activity

INTERVENTIONS:
Behavioral: Standard of Care advice on physical activity — Oral advice on exercise from a physician.
  Arms: Standard of care
Behavioral: Structured advice on physical activity — A leaflet with instructions and images on different forms of physical activities as well as clear recommendations on when to perform these.
  Arms: Active intervention

SUMMARY:
The study will compare two forms of advice regarding physical activity for patients hospitalized with cirrhosis that are preparing for leaving the hospital. One arm consists of current standard of care: simple oral advice on exercise. One arm instead gives patients a structured but simple paper template on physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis diagnosed with previous clinical assessment and radiology (de-formed liver, noduli, varices, collaterals, splenomegaly >12 cm) or with biopsy (fibrosis grade 4). ICD-code K70.3, K74.6.
* MELD < 25
* Understanding the Swedish language.
* Signed informed consent.

Exclusion Criteria:

* Performance status ≥3.
* Severe pain which prevents the patient to perform the physical activities, as judged by the attending physician at time of discharge.
* Previously liver transplanted
* Unlikely to be compliant to follow-up (living in other parts of Sweden), as judged by the attending physician at time of discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life summary score, as measured with the CLDQ tool | 3 months
  Change in quality of life, as measured with the CLDQ tool (gives a summary score between 1-7, a higher score suggests a better quality of life).

SECONDARY OUTCOMES:
Frailty | 3 months
  Frailty as measured with the Liver Frailty Index.
MELD | 3 months
  Model of End-stage Liver Disease score (range 6-40, a higher score indicates a worse prognosis)
Mortality | 3 months
  Overall mortality

CONTACTS AND LOCATIONS:
Overall Officials: Hannes Hagström, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No